CLINICAL TRIAL: NCT04543591
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Ravulizumab in Adult and Adolescent Participants Who Have Thrombotic Microangiopathy (TMA) After Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Ravulizumab in Thrombotic Microangiopathy After Hematopoietic Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN1210-TMA-313
Record Dates: First submitted 2020-08-17; First posted 2020-09-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thrombotic Microangiopathy
Keywords: Thrombotic Microangiopathy (TMA) Ultomiris; Ravulizumab; Hematopoietic Stem Cell Transplant (HSCT) Transplant-associated TMA; HSCT-TMA
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): In Stage 1, all participants will receive open-label ravulizumab plus Best Supportive Care (BSC).
  In Stage 2, participants will receive blinded ravulizumab plus Best Supportive Care (BSC).
  Interventions: Biological: Ravulizumab; Other: Best supportive care
- Placebo (Placebo Comparator): In Stage 2, participants randomized to the placebo arm will receive matching placebo plus BSC.
  Interventions: Other: Placebo; Other: Best supportive care

INTERVENTIONS:
Biological: Ravulizumab — Weight-based doses of ravulizumab will be administered intravenously as loading dose regimen followed by maintenance dosing every 8 weeks.
  Other Names: Ultomiris, ALXN1210
  Arms: Ravulizumab
Other: Placebo — Matching placebo
  Arms: Placebo
Other: Best supportive care — Participants will receive medications, therapies, and interventions per standard hospital treatment protocols (unless specifically prohibited by the protocol).

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of ravulizumab in adult and adolescent participants with hematopoietic stem cell transplant-associated thrombotic microangiopathy (HSCT-TMA). In Stage 1, an open-label, single-arm period, the dosing regimen will be confirmed. In Stage 2, participants will be randomized to receive either blinded ravulizumab plus best supportive care or matching placebo plus best supportive care. The treatment period is 26 weeks (open-label for Stage 1, and randomized, double-blind, and placebo-controlled for Stage 2) followed by a 26-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years of age or older at time of consent/assent.
2. Received HSCT within the past 12 months.
3. Diagnosis of TMA that persists for at least 72 hours after initial management of any triggering agent/condition.
4. A TMA diagnosis based on meeting the laboratory-based criteria during the Screening Period and/or ≤14 days prior to the Screening Period.
5. Body weight ≥ 30 kilograms at Screening or ≤7 days prior to the start of the Screening Period (date of consent).
6. Female participants of childbearing potential and male participants with female partners of childbearing potential must use highly effective contraception.
7. Participants must be vaccinated against meningococcal infections if clinically feasible. Participants who cannot receive meningococcal vaccine should receive antibiotic prophylaxis. Participants <18 years of age must be re-vaccinated against Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae if clinically feasible.
8. Participants or their legally authorized representative must be capable of giving signed informed consent or assent.

Exclusion Criteria:

1. Thrombotic thrombocytopenic purpura (TTP) evidenced by ADAMTS13 deficiency
2. Known Shiga toxin-related hemolytic uremic syndrome as demonstrated by positive test.
3. Positive direct Coombs test indicative of a clinically significant immune-mediated hemolysis not due to TMA.
4. Clinical diagnosis of disseminated intravascular coagulation (DIC).
5. Known bone marrow/graft failure for the current HSCT.
6. Diagnosis of veno-occlusive disease which is unresolved at the time of Screening.
7. Human immunodeficiency virus (HIV) infection.
8. Unresolved meningococcal disease.
9. Presence of sepsis requiring vasopressor support.
10. Pregnancy or breastfeeding.
11. Hypersensitivity to murine proteins or to one of the excipients of ravulizumab.
12. Any ongoing or history of medical or psychological conditions unrelated to HSCT-TMA that could increase the risk to the participant or confound the outcome of the study.
13. Respiratory failure requiring mechanical ventilation.
14. Acute and/or chronic heart failure with an ejection fraction ≤ 40%.
15. Previously or currently treated with a complement inhibitor.
16. Participation in an interventional treatment study of any therapy for TMA.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 26 weeks (treatment period)
  Event free survival during the 26 weeks treatment period defined as the time from randomization until the first of the two following events: death and clinical worsening.

SECONDARY OUTCOMES:
Time To TMA Response | 26 weeks (treatment period)
Change from Baseline in eGFR | 26 weeks (treatment period) and 52 weeks
Overall Survival | Day 100, 26 weeks (treatment period), and 52 weeks
Non-relapse Mortality | Day 100, 26 weeks (treatment period), and 52 weeks
Hematologic Response | 26 weeks (treatment period)
TMA response and time to response for each individual component of TMA | 26 weeks (treatment period)
Time to Hematologic Response | 26 weeks (treatment period)
Hemoglobin Response | 26 weeks (treatment period)
Partial Response | 26 weeks (treatment period)
Loss of TMA Response | 26 weeks (treatment period)
Duration of TMA Response | 26 weeks (treatment period) and 52 weeks
Changes from Baseline in Haptoglobin, Platelets, LDH, and Hemoglobin | 26 weeks (treatment period) and 52 weeks
Modified TMA Response | 26 weeks (treatment period)
Change from baseline in TMA-associated organ dysfunction in renal system, cardiovascular system, pulmonary system, CNS, and GI system | 26 weeks (treatment period) and 52 weeks
TMA Relapse | Follow-up Period
Platelet Response | 26 weeks (treatment period)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (5):
  - Research Site, Tampa, Florida
  - Research Site, Grosse Pointe Farms, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Seattle, Washington
- Research Site, Parkville, Australia
- Belgium (4):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Chênée
  - Research Site, Yvoir
- Brazil (7):
  - Research Site, Cerqueira César
  - Research Site, Florianópolis
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Research Site, Calgary, Alberta, Canada
- China (2):
  - Research Site, Suzhou
  - Research Site, Tianjin
- France (3):
  - Research Site, Angers
  - Research Site, La Tronche
  - Research Site, Nice
- Germany (2):
  - Research Site, Hamburg
  - Research Site, Ulm
- Greece (3):
  - Research Site, Athens
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Israel (2):
  - Research Site, Halfa
  - Research Site, Ramat Gan
- Italy (2):
  - Research Site, Roma
  - Research Site, Udine
- Japan (14):
  - Research Site, Akita
  - Research Site, Anjo
  - Research Site, Chiba
  - Research Site, Fukushima
  - Research Site, Isehara-shi
  - Research Site, Kurashiki-shi
  - Research Site, Minatoku
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Suita-shi
  - Research Site, Tsukuba
  - Research Site, Wakayama
- Research Site, Groningen, Netherlands
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Seville
- Research Site, Huddinge, Sweden
- United Kingdom (2):
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: No